CLINICAL TRIAL: NCT01629602
Title: Treatment of Soft Tissue Loss With Nerve Defect in the Finger Using the Boomerang Nerve Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TSChen4112
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2011-05

CONDITIONS: Soft Tissue Loss With Nerve Defect
Keywords: defect;; dorsal branch of the proper digital nerve;; proper digital nerve;; vascularized nerve graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- vascularized nerve graft (Experimental): The investigators combined the nerve branch with the boomerang flap for simultaneous repair of soft tissue loss and PDN defect in these awkward areas.
  Interventions: Procedure: the Boomerang Nerve Flap

INTERVENTIONS:
Procedure: the Boomerang Nerve Flap — The nerve branch was combined with the boomerang flap for simultaneous repair of soft tissue loss and PDN defect in these awkward areas.

SUMMARY:
Soft tissue loss with proper digital nerve (PDN) defect in the finger results in sensory loss of the finger pulp. Reconstruction of these complex soft tissue defects continues to be a challenge problem. To resolve this problem, we combined the nerve branch with the boomerang flap for simultaneous repair of soft tissue loss and PDN defect in these awkward areas. For comparison, we also collected a consecutive series of 32 patients with similar injury in the finger treated using a cross finger flap and a secondary free nerve graft.

DETAILED DESCRIPTION:
The patients in this study group were required to meet all of the following criteria: soft tissue loss between the midpoint of the distal phalanx and PIP joint; associated PDN defect 1 to 4 cm in length; single or double PDN defects; and simultaneous repair of soft tissue loss and PDN defect. Patients were excluded when they had the following: injury to the course of the vascular pedicle or the donor site or the donor nerve; PDN defect less than 1 cm or larger than 4 cm in length; direct PDN repair; and thumb neurocutaneous defects.

ELIGIBILITY:
Inclusion Criteria:

* soft tissue loss between the midpoint of the distal phalanx and PIP joint; - associated PDN defect 1 to 4 cm in length;
* single or double PDN defects;
* simultaneous repair of soft tissue loss and PDN defect.

Exclusion Criteria:

* injury to the course of the vascular pedicle or the donor nerve;
* PDN defect less than 1 cm or larger than 4 cm in length;
* direct PDN repair;
* thumb neurocutaneous defects.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination test | from 18 to 24 months
  The test points were at the centers of the radial and ulnar portions of the finger pulp, the flap and the donor sites separately.

SECONDARY OUTCOMES:
Cold Intolerance Severity Score (CISS) questionnaire | from 18 to 24 months
  The maximum score was 100 and was grouped into mild (0-25), moderate (26-50), severe (51-75) and extreme severity (76-100).

REFERENCES:
- [Derived] Chen C, Tang P, Zhang X. Treatment of soft-tissue loss with nerve defect in the finger using the boomerang nerve flap. Plast Reconstr Surg. 2013 Jan;131(1):44e-54e. doi: 10.1097/PRS.0b013e3182729f5e. PMID 23271553